CLINICAL TRIAL: NCT05569512
Title: A Phase 1/2 Trial of Uproleselan Combined With High Dose Busulfan Pre-Transplant Conditioning in Hematopoietic Stem Cell Transplantation for Patients With Chemotherapy Resistant Acute Myeloid Leukemia
Brief Title: Uproleselan With Pre-Transplant Conditioning in Hematopoietic Stem Cell Transplantation for AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: On 7/26/24 the Sponsor-Investigator was notified GlycoMimetics was terminating contracting for NCT05569512 following company restructuring. This notification came ahead of the study meeting criteria to progress from Phase 1 to Phase 2.
Sponsor: Malika Kapadia (Other)
Collaborators: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Malika Kapadia, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-063
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia; Pediatric Cancer
Keywords: Acute Myeloid Leukemia; Pediatric Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — uproleselan; fludarabine; fludarabine phosphate; Clofarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Uproleselan with pre-transplant conditioning (Experimental): Participants will receive IV uproleselan on day -8 prior to stem cell transplant. Uproleselan will be administered IV twice daily from day -7 through day -2.
  Participants will also receive a standard pre-transplant conditioning regimen with fludarabine, clofarabine and busulfan. Each of these 3 drugs will be administered IV once daily from day -7 through day -4.
  Interventions: Drug: Uproleselan; Drug: Fludarabine; Drug: Clofarabine; Drug: Busulfan

INTERVENTIONS:
Drug: Uproleselan — Administered by intravenous infusion
Drug: Fludarabine — Administered by intravenous infusion
  Other Names: Fludara
Drug: Clofarabine — Administered by intravenous infusion
  Other Names: Clolar
Drug: Busulfan — Administered by intravenous infusion
  Other Names: Busulfex; Myleran

SUMMARY:
This research study is studying a new drug, uproleselan, to see if it is safe and effective in decreasing relapse after stem cell transplant and improving leukemia-free survival in pediatric patients with acute myeloid leukemia (AML).

The name of the study drugs involved in this study are:

* Uproleselan
* Busulfan
* Clofarabine
* Fludarabine
* Tacrolimus
* Methotrexate
* Mycophenolate Mofetil

DETAILED DESCRIPTION:
This is a single arm, multi-center, phase 1/2 trial involving the use of the study drug, uproleselan, as part of the pre stem cell transplant conditioning regimen for pediatric patients with acute myeloid leukemia (AML). This study is looking to learn what dose of uproleselan should be given and the safety of uproleselan when combined with other drugs as part of the pre stem cell transplant conditioning regimen.

The U.S. Food and Drug Administration (FDA) has not approved uproleselan as a treatment for any disease. This is the first time that uproleselan will be given to children. Uproleselan is expected to treat acute myeloid leukemia (AML) by making AML cells sensitive to chemotherapy drugs that are part of standard of care pre-transplant conditioning regimen which could help make the transplant more effective..The standard of care conditioning regimen will include the drugs busulfan, clofarabine, and fludarabine. The standard of care drugs tacrolimus, and either methotrexate or mycophenolate mofetil will be used during the stem cell transplant course.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive study drug doses for 7 days before their stem cell transplant and will be followed for 2 years following their stem cell transplant.

It is expected that about 28 people will take part in this research study.

GlycoMimetics, Inc., a pharmaceutical company, is supporting this research study by providing the study drug (uproleselan) and funding for some of the laboratory tests.

On 7/26/24 the Sponsor-Investigator was notified GlycoMimetics, Inc. was terminating contracting for NCT05569512 following company restructuring. One subject was enrolled on the study prior to termination. The study did not proceed from Phase 1 to Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 months and ≤ 39 years

  * The minimum and maximum number of subjects enrolled on the study are 20 and 28, respectively. In order to ensure at least 70% of the population are under the age of 18 years of age, the number of subjects >=18 years old will be limited as follows:
  * At least 7 of the first 10 subjects must be under 18 years old
  * At least 7 of the second 10 subjects must be under 18 years old
  * At least 6 of the last 8 subjects enrolled must be under 18 years old
* Lansky/Karnofsky performance status ≥70% (see Appendix A)
* Weight ≥10 kg
* Acute myeloid leukemia that arises de novo or is secondary to:

  * cytotoxic chemoradiotherapy
  * myelodysplastic syndrome
  * a leukemia predisposition syndrome or inherited marrow failure syndrome other than ones associated with transplant-related morbidity and mortality. A predisposition resulting from a germline RUNX1 mutation is example of an eligible disorder. Fanconi Anemia and Dyskeratosis Congenita are examples of ineligible disorders.
* Disease status: Multidimensional flow cytometry (MDF) to assess disease status for eligibility will be performed centrally by Hematologics.

  * In a first or second complete remission (defined as marrow with ≤1% leukemic blasts by MDF and no evidence of extramedullary disease) with minimal residual disease (MRD, defined as marrow with ≥0.05% leukemic blasts by MDF) after at least 2 cycles of induction/re-induction chemotherapy.
  * Have newly diagnosed disease or disease in first relapse that is refractory (defined as marrow with >1% leukemic blasts by MDF or persistence of extramedullary disease) to at least 2 cycles of induction/re-induction chemotherapy.

This sample will be used for eligibility as well as correlative biomarkers. Please see section 9.2 for details regarding collection, processing, and shipping of the sample.

* Graft and Donor Types:

  * Patients must be receiving bone marrow or peripheral blood stem cells from a HLA identical related or HLA matched unrelated (allele level matched at A, B, C and DRB1 loci) donor.
  * Eligibility of prospective donors should be determined in compliance with requirements of 21 CFR Part 1271. This should include donor screening for COVID-19 exposure or infection. https://www.fda.gov/vaccines-blood-biologics/safety-availability-biologics/updated-information-human-cell-tissue-or-cellular-or-tissue-based-product-hctp-establishments
* Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had a previous hematopoietic stem cell transplantation
* Participants who have had prior treatment with uproleselan
* CNS 3 disease at time of admission for HSCT. Patients previously diagnosed CNS 3 disease that has improved (CNS1 or CNS2) will be eligible. (See Section 3.3 for definitions).
* Down Syndrome
* Fanconi Anemia, Dyskeratosis Congenita and other disorders associated with excess risk for transplant related toxicities
* Acute Promyelocytic Leukemia
* Multiply relapsed (≥2) disease
* Pregnancy (positive serum beta-HCG) or breastfeeding Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with uproleselan, breastfeeding should be discontinued if the mother is treated with uproleselan. These potential risks also apply to other agents used in this study.
* Absolute neutrophil count <300/μL due to treatment (chemotherapy or immunotherapy).

Patients with neutropenia due to disease related marrow dysfunction (refractory disease, underlying myelodysplasia or an underlying marrow failure disorder) will be eligible regardless of the absolute neutrophil count. However, enrolling centers must provide clear evidence that the neutrophil count is not rising, that the patient does not have an inadequately controlled infection (see section 3.2.15), and that the patient is on broad anti-fungal prophylaxis. Given the serious risk associated with starting conditioning in patients with severe neutropenia, centers are encouraged to delay transplant if they have any reason to believe that the absolute neutrophil count may improve.

* Estimated GFR of <60 mL/min/1.73 m2. Estimated GFR may be calculated using the CKD-EPI Creatinine Equation (2009) for patients ≥19 years or creatinine-based Bedside Schwartz equation (2009) for patients <19 years. It is recommended that estimates be determined using the calculators found on the National Kidney Foundation website. the (https://www.kidney.org/professionals/KDOQI/gfr_calculator). Any patient for whom these equations yields a GFR less than 90 mL/min/1.73 m2 should have radionucleotide testing. Measurement of 24-hour urine creatinine clearance is not an acceptable substitute for radionucleotide testing.
* Cardiac ejection fraction <50% or shortening fraction <27%
* Total bilirubin (with elevated direct bilirubin) or ALT >2 X ULN.
* Pulmonary disease with FVC, FEV1 or DLCO (corrected for hemoglobin) <50 % predicted or requiring supplemental oxygen. Children who are developmentally unable to perform pulmonary function testing will be assessed solely on their need for supplemental oxygen
* Active hepatitis B or C infection
* Active, poorly controlled infections. In patients being treated for infection at the time of enrollment, source documentation of the results of all microbiologic, radiographic and pathology assessments performed for diagnosis and for evaluation of response to treatment will be required.
* Patients with a known history of HIV are excluded, unless they meet all of the following conditions:

  * No history of HIV complications with the exception of CD4 count <200 cells/mm3
  * No antiretroviral therapy with overlapping toxicity such as myelosuppression
  * CD4 count >500 cells/mm3 prior to the diagnosis of relapsed AML
  * HIV viral loads below the limit of detection
  * No history of highly active antiretroviral therapy (HAART)-resistant HIV
* Patients who have received another investigational drug within 28 days or 5 half-lives (whichever is longer).

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Recommend Phase 2 Dose | Day -8 pre- transplant through post-transplant Day +30
  Dose recommended by study team based on maximum tolerated dose (MTD). Highest dose level at or below the maximally administered dose where ≤1 out of 6 patients experienced a Dose Limiting Toxicity (DLT)
Dose Limiting Toxicity (DLT) Phase 1 | Transplant Day 0 through post-transplant Day +30
  All observed toxicities will be summarized using frequencies, proportions, and 95% confidence intervals by type (organ affected or laboratory determination), severity (by CTCAEv5.0), attribution, and expectedness. Only the maximum grade for each type of toxicity will be tabulated for each patient.
Dose Limiting Toxicity (DLT) Phase 2 | Transplant Day 0 through post-transplant Day +30
  All observed toxicities will be summarized using frequencies, proportions, and 95% confidence intervals by type (organ affected or laboratory determination), severity (by CTCAEv5.0), attribution, and expectedness. Only the maximum grade for each type of toxicity will be tabulated for each patient.

SECONDARY OUTCOMES:
Uproleselan Pharmacokinetics | Day -8 pre-transplant to day -4 pre- transplant
  Blood samples will be drawn for measurement of uproleselan plasma levels with the day -8 dose and the first day -4 dose. Four 1 ml samples will be drawn each day for patients less than 6 years. Five 2 ml samples will be drawn each day for patients 6 years and older. Measurements will be used to estimate uproleselan area under the curve.
12-month Leukemia-Free Survival (LFS) | 12 months
  Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria:
Overall Survival (OS) | Date of transplant (Day 0) to 2 years post stem cell transplant
  Overall Survival (OS) is based on the Kaplan-Meier method and defined as the time from study entry to death or censored at date last known alive per immune RECIST (iRECIST)
Relapse Rate at the RP2D | Up to 2 years
  Rate of Relapse defined as the proportion of patients that has relapse on treatment or during the follow-up period
Number of Patients with Severe Oral or Gastrointestinal Mucositis | Between day 0 and post-transplant day 14
  Defined as all grade 3 or higher oral or gastrointestinal mucositis related adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5.

CONTACTS AND LOCATIONS:
Overall Officials: Malika Kapadia, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Helen DeVos Children's Hospital/Spectrum Health, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu

DOCUMENTS (1):
  • Study Protocol (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT05569512/Prot_000.pdf